CLINICAL TRIAL: NCT02844413
Title: The Influence of Regular Aerobic Interval Training on Blood Pressure and Arterial Stiffness Amongst Hypertensive Subjects
Brief Title: Physical Exercises Influence on Blood Pressure and Arterial Stiffness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Kameczura, MD, PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMUJ-2015/67
Record Dates: First submitted 2016-07-12; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): implementation of aerobic interval training
  Interventions: Other: aerobic interval training
- control group (No Intervention): control group

INTERVENTIONS:
Other: aerobic interval training — In the first group (G1), aerobic interval training (AIT) was undertaken for 5 months (40 professional AIT sessions performed two times per week in 50 minute sessions) and followed a specially developed program. The second control group (G2), did not attend any training sessions but received medical advice on how to maintain physical activity as outlined by JNC hypertension guidelines
  Other Names: AIT
  Arms: study group

SUMMARY:
Regular exercise is recommended as an adjuvant treatment in hypertensive subjects by both European and American guidelines. Crucially, however, there are no precise recommendations on the type of physical exercise and how it should be instituted A relatively short period (5 months) of regular aerobic interval training (AIT), significantly decreased blood pressure, pulse wave velocity, and most applanation tonometry indexes in hypertensive subjects also undertaking pharmacological treatment in our study.

DETAILED DESCRIPTION:
Regular physical exercise appears to potentiate the effects of pharmacological treatment for arterial hypertension. As such, regular exercise is recommended as an adjuvant treatment in hypertensive subjects by both European and American guidelines. Crucially, however, there are no precise recommendations on the type of physical exercise and how it should be instituted. Aerobic Interval Training (AIT) is a new and novel type training that appears to be beneficial to patients suffering from various medical conditions. There is a distinct lack of evidence on how it affects arterial hypertension. The aim of this study was to evaluate the influence of a 5 month period of regular AIT on blood pressure, carotid femoral pulse wave velocity (PWV) and applanation tonometry indexes in patients previously treated pharmacologically for mild or moderate arterial hypertension.

The study group consisted of 60 hypertensive subjects (30 males, 30 females) (age 54.45 ± 8.52 years) who had previously undergone at least 2 years of combined anti-hypertensive therapy and who had well controlled hypertension, i.e. below 140/90 mmHg. Their pharmacological treatment did not change during the study period. The study group was randomly divided into 2 subgroups. In the first group (G1), AIT was undertaken for 5 months (40 professional AIT sessions performed two times per week in 50 minute sessions) and followed a specially developed program. The second control group (G2), did not attend any training sessions but received medical advice on how to maintain physical activity as outlined by JNC (Joint National Committee) hypertension guidelines. During the baseline visit and then at five months (final visit), both groups underwent testing for office BP (blood pressure), PWV and applanation tonometry indexes using the SphygmoCor® device and the Complior® device.

ELIGIBILITY:
Inclusion Criteria:

* subjects who have had previously undergone at least 2 years of combined antihypertensive therapy and who had well controlled hypertension, i.e. below 140/90 mmHg
* subjects whos pharmacological treatment did not change during the study period

Exclusion Criteria:

* Secondary hypertension
* Chronic kidney or liver failure
* Grade 3 hypertension as defined by European Society of Hypertension 2013
* Chronic obstructive pulmonary disease
* The need for the use of 3 antihypertensives
* Diabetes or other illness affected carbohydrate metabolism
* Previous myocardial infarction
* Other serious conditions which might shorten survival time
* Previous stroke or transient ichemic attack (TIA)
* Other conditions affecting the locomotor system which would significantly limit the ability to undertake exercise
* Symptomatic heart failure
* Lack of informed consent

Ages: 51 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity augmentation of 1.04 [m/s] | 5 months

SECONDARY OUTCOMES:
systolic blood pressure reduction of 3.9 [mmHg] and diastolic blood pressure reduction of 2.7 [mmHg] | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Kameczura, MD, PhD, Principal Investigator — Jagiellonian University

IPD SHARING:
Plan to Share IPD: Undecided